CLINICAL TRIAL: NCT00961051
Title: Evaluation of an Investigational MPS
Brief Title: Evaluation of an Investigational Multi-Purpose Solution (MPS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: COBR-105-9608
Record Dates: First submitted 2009-07-27; First posted 2009-08-18 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2013-12

CONDITIONS: Study Focus is Healthy Contact Lens Wearers
Keywords: adapted contact lens wearers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational MPS (Experimental): Investigational multipurpose disinfecting solution (study MPS)
  Interventions: Device: Investigational MPS
- Predicate MPS (Active Comparator): Opti-Free RepleniSH multipurpose disinfecting solution (predicate MPS)
  Interventions: Device: Opti-Free

INTERVENTIONS:
Device: Investigational MPS — Multi-purpose solution
  Other Names: Cobra
  Arms: Investigational MPS
Device: Opti-Free — Multi-purpose solution
  Other Names: RepleniSH
  Arms: Predicate MPS

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an investigational multi-purpose contact lens solution.

DETAILED DESCRIPTION:
A new multi-purpose solution has been developed for optimal lens disinfection and lens wearing comfort, compatible with a wide variety of commercially available lenses. Ten investigative sites were selected to evaluate 274 soft contact lens wearers in a parallel group study of one investigational multi-purpose solution and one marketed predicate solution.

ELIGIBILITY:
Inclusion Criteria:

* Have successfully worn hydrogel contact lenses of the same material to be worn during the study
* Have normal eyes (with the exception of unaided visual acuity)
* Have successfully used a multi-purpose contact lens care solution
* Have acceptable visual acuity and lens wearing comfort at time of enrollment

Exclusion Criteria:

* Concurrently enrolled another clinical trial
* Have a known sensitivity to any study product ingredient(s)
* Have a condition that may put them at significant risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Tarantino, OD, Study Chair — Abbott Medical Optics
Locations (9):
- United States (9):
  - Complete Family Vision Center, San Diego, California
  - Eye Care Associates of Hawaii, Waipahu, Hawaii
  - Insight Eyecare, Warrensburg, Missouri
  - Drs. Quinn, Quinn & Associates, Athens, Ohio
  - Western Reserve Vision Care, Beachwood, Ohio
  - Central Ohio Eyecare, Columbus, Ohio
  - Northeastern Eye Institute, Scranton, Pennsylvania
  - West Bay Eye Associates, Warwick, Rhode Island
  - Ziegler Leffingwell Eyecare, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for this study were chosen from the normal hydrogel contact lens-wearing patient populations at each of the investigational sites according to the following inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Investigational MPS | Predicate MPS
Started | 177 | 93
Completed | 165 | 79
Not Completed | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational MPS | Predicate MPS | Total
Number analyzed (Participants) | 177 | 93 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 177 | 93 | 270
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 65 | 183
  Male | 59 | 28 | 87
Region of Enrollment [Number; unit: participants]
  United States | 177 | 93 | 270

OUTCOME MEASURES:

1. Primary Outcome: Mean Lens Cleanliness as Measured by Light Reflectance
Description: Lens cleanliness was assessed by total light reflectance, which is a computerized quantitative assessment conducted in a laboratory. The amount of light that scattered off the lens surface in a light field and was assessed using a light reflectance score that ranged from 0 (maximum lens cleanliness; clean/clear) to100 (minimum lens cleanliness; dirty/opaque).
Time Frame: Day 30
Population: Lens cleanliness analysis could only be done on subjects whose lenses were returned for analysis. Out of 270 subjects, 253 returned their study lenses to the sponsor for lab analysis (169 + 84 = 253).
Measure: Mean (Standard Deviation); unit: light reflectance score
Arm/Group | Investigational MPS | Predicate MPS
Number analyzed (Participants) | 169 | 84
light reflectance score | 65.5 (13.92) | 66.8 (14.95)

2. Secondary Outcome: Number of Subjects With no Corneal Staining
Description: Corneal staining was performed via slit lamp observation of the corneal through a cobalt blue filter and a yellow #12 or #15 filter Wratten filter following contact lens removal and installation of standard sodium fluorescein.
Time Frame: Day 180
Measure: Number; unit: participants
Arm/Group | Investigational MPS | Predicate MPS
Number analyzed (Participants) | 165 | 79
participants | 129 | 64

ADVERSE EVENTS:
Arm/Group | Investigational MPS | Predicate MPS
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/93
Other Adverse Events (participants affected / at risk) | 6/177 | 12/93
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational MPS (N=177) | Predicate MPS (N=93)
Red eye (Eye disorders) | 1 (1) | 2 (2)
Conjunctivitis (Eye disorders) | 2 (2) | 1 (1)
Corneal infiltrates (Eye disorders) | 1 (1) | 0 (0)
Corneal ulcer (Eye disorders) | 1 (1) | 0 (0)
Foreign body sensation (Eye disorders) | 1 (1) | 0 (0)
Seasonal eye allergies (Eye disorders) | 0 (0) | 2 (2) — Seasonal eye allergies may also cause dry eyes, redness, blurry vision, and light sensitivity
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Superficial punctate keratopathy (Eye disorders) | 0 (0) | 1 (1)
Giant papillary conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Recurrent corneal erosion (Eye disorders) | 0 (0) | 1 (1)
Hypersensitivity to study solution (Eye disorders) | 0 (0) | 2 (2)
Hordeolum (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to publication release and can embargo communications regarding trials results for a period that is more than 90 days but less than or equal to 18 months from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.